CLINICAL TRIAL: NCT01849289
Title: A Trial Comparing Efficacy and Safety of Insulin Degludec and Insulin Glargine in Insulin naïve Subjects With Type 2 Diabetes (BEGIN™: ONCE)
Brief Title: A Trial Comparing Efficacy and Safety of Insulin Degludec and Insulin Glargine in Insulin naïve Subjects With Type 2 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3587; U1111-1121-5325 (Other: WHO)
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Degludec (Experimental)
  Interventions: Drug: Insulin Degludec
- Insulin Glargine (Experimental)
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Degludec — Administered subcutaneously (under the skin), dose individually adjusted, once daily in combination with metformin at the unchanged, stable, pre-randomisation dose level and dosing frequency.
  Other Names: NN1250
  Arms: Insulin Degludec
Drug: Insulin Glargine — Administered subcutaneously (under the skin), dose individually adjusted, once daily in combination with metformin at the unchanged, stable, pre-randomisation dose level and dosing frequency.
  Arms: Insulin Glargine

SUMMARY:
This trial was conducted in Africa, Asia, Europe, North and South America. The aim of the trial was to compare efficacy and safety of insulin degludec and insulin glargine in insulin naïve subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed clinically) for at least 6 months
* Insulin naïve subjects (Allowed are: previous short term insulin treatment up to 14 days; treatment during hospitalisation or during gestational diabetes is allowed for periods longer than 14 days)
* Current treatment: metformin monotherapy or metformin in any combination with an insulin secretagogue (sulfonylurea or glinide), dipeptidyl peptidase IV (DPP-IV) inhibitor, alfa-glucosidase-inhibitors (acarbose) with unchanged dosing for at least 3 months prior to randomisation (Visit 2) with the minimum doses stated: metformin: alone or in combination (including fixed combination) 1500 mg daily, or maximum tolerated dose (at least 1000 mg daily), insulin secretagogue (sulfonylurea or glinide): minimum half of the daily maximal dose according to local labelling, DPP-IV inhibitor: minimum 100 mg daily or according to local labelling, alfa-glucosidase-inhibitors (acarbose): minimum half of the daily maximal dose or maximum tolerated dose
* HbA1c (glycosylated haemoglobin) 7.0-10.0% (both inclusive) by central laboratory analysis
* BMI (Body Mass Index) below or equal to 40.0 kg/m^2

Exclusion Criteria:

* Treatment with TZDs (thiazoledinedione), or GLP-1 (glucagon-like peptide 1) receptor agonists within the last 3 months prior to Visit 1 (screening)
* Anticipated change in concomitant medication known to interfere significantly with glucose metabolism, such as systemic corticosteroids, beta-blockers, MAO (monoamine oxidase) inhibitors
* Cardiovascular disease within the last 6 months prior to Visit 1 (screening) defined as stroke; decompensated heart failure NYHA (New York Heart Association) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Any clinically significant disease or disorder, except for conditions associated with type 2 diabetes mellitus, which in the Investigator's opinion could interfere with the results of the trial
* Previous participation in this trial. Participation is defined as randomised. Re-screening of screening failures is allowed only once within the limits of the recruitment period
* Known or suspected hypersensitivity to trial product(s) or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2013-06-02 (Actual); Primary Completion 2014-05-15 (Actual); Study Completion 2014-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (66):
- United States (18):
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Crestview Hills, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, Simpsonville, South Carolina
  - Novo Nordisk Investigational Site, Jackson, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
- Brazil (3):
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Porto Alegre
  - Novo Nordisk Investigational Site, São Paulo
- Canada (11):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Burnaby, British Columbia
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Victoria, British Columbia
  - Novo Nordisk Investigational Site, Burlington, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Newmarket, Ontario
  - Novo Nordisk Investigational Site, Sarnia, Ontario
  - Novo Nordisk Investigational Site, Strathroy, Ontario
  - Novo Nordisk Investigational Site, Québec, Quebec
  - Novo Nordisk Investigational Site, Trois-Rivières, Quebec
- China (22):
  - Novo Nordisk Investigational Site, Hefei, Anhui
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Fuzhou, Fujian
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Nanning, Guangxi
  - Novo Nordisk Investigational Site, Guiyang, Guizhou
  - Novo Nordisk Investigational Site, Shijiazhuang, Hebei
  - Novo Nordisk Investigational Site, Harbin, Heilongjiang
  - Novo Nordisk Investigational Site, Wuhan, Hubei
  - Novo Nordisk Investigational Site, Yueyang, Hunan
  - Novo Nordisk Investigational Site, Yangzhou, Jiangsu
  - Novo Nordisk Investigational Site, Zhenjiang, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Changchun, Jilin
  - Novo Nordisk Investigational Site, Siping, Jilin
  - Novo Nordisk Investigational Site, Shenyang, Liaoning
  - Novo Nordisk Investigational Site, Xi'an, Shaanxi
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Kunming, Yunnan
  - Novo Nordisk Investigational Site, Hangzhou, Zhejiang
  - Novo Nordisk Investigational Site, Wenzhou, Zhejiang
- Romania (5):
  - Novo Nordisk Investigational Site, Oradea, Bihor County
  - Novo Nordisk Investigational Site, Buzău, Buzău
  - Novo Nordisk Investigational Site, Sibiu, Sibiu County
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Galati
- South Africa (3):
  - Novo Nordisk Investigational Site, George, Eastern Cape
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
- Ukraine (4):
  - Novo Nordisk Investigational Site, Dnipro
  - Novo Nordisk Investigational Site, Kiev
  - Novo Nordisk Investigational Site, Mykolaiv
  - Novo Nordisk Investigational Site, Vinnitsa

REFERENCES:
- [Result] Pan C, Gross JL, Yang W, Lv X, Sun L, Hansen CT, Xu H, Wagner R. A Multinational, Randomized, Open-label, Treat-to-Target Trial Comparing Insulin Degludec and Insulin Glargine in Insulin-Naive Patients with Type 2 Diabetes Mellitus. Drugs R D. 2016 Jun;16(2):239-49. doi: 10.1007/s40268-016-0134-z. PMID 27098525
- [Derived] Mu YM, Guo LX, Li L, Li YM, Xu XJ, Li QM, Xu MT, Zhu LY, Yuan GY, Liu Y, Xu C, Wang ZJ, Shen FX, Luo Y, Liu JY, Li QF, Wang WH, Lai XY, Xu HF, Pan CY. [The efficacy and safety of insulin degludec versus insulin glargine in insulin-naive subjects with type 2 diabetes: results of a Chinese cohort from a multinational randomized controlled trial]. Zhonghua Nei Ke Za Zhi. 2017 Sep 1;56(9):660-666. doi: 10.3760/cma.j.issn.0578-1426.2017.09.008. Chinese. PMID 28870034
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 68 sites in six countries as follows:
  Brazil: 3 sites; Canada: 7 sites; China: 37 sites; South Africa: 4 sites; Ukraine: 6 sites; United States: 11 sites.
Pre-assignment Details: The subjects discontinued their current Oral Antidiabetic drug (OAD) treatment at Visit 2 (randomisation visit) except for metformin, before starting the treatment with trial drugs.
Groups:
- IDeg OD: Insulin degludec (IDeg) 10U was injected subcutaneously (under the skin) once daily (OD) in the evening (start of main evening meal to bedtime) either in the thigh, upper arm (deltoid area) or abdomen along with metformin given orally for 26 weeks. At last treatment visit (Visit 28) subjects were instructed to switch basal insulin treatment to the intermediate acting insulin NPH until the follow-up visit (Visit 29).
- IGlar OD: Insulin glargine (IGlar) 10U was injected subcutaneously (under the skin) once daily (OD) in the evening (start of main evening meal to bedtime) either in the thigh, upper arm (deltoid area) or abdomen along with metformin given orally for 26 weeks. At last treatment visit (Visit 28) subjects were instructed to switch basal insulin treatment to the intermediate acting insulin NPH until the follow-up visit (Visit 29).
Period: Overall Study
Arm/Group | IDeg OD | IGlar OD
Started | 555 | 278
Exposed | 553 (2 subjects withdrew prior to exposure of trial products) | 278
Completed | 523 | 254
Not Completed | 32 | 24
Not completed — Adverse Event | 3 | 3
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal criteria | 1 | 0
Not completed — Unclassified | 25 | 18

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg OD | IGlar OD | Total
Number analyzed (Participants) | 555 | 278 | 833
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.7) | 56.6 (9.2) | 56.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 256 | 146 | 402
  Male | 299 | 132 | 431
HbA1c [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.9) | 8.3 (0.8) | 8.3 (0.8)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.4 (2.4) | 9.4 (2.5) | 9.4 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (%) (Analysed by Central Laboratory)
Description: Change from baseline in HbA1c (%) after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects. Last Observation Carried Forward (LOCF) values were presented for this endpoint.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 555 | 278
percentage of glycosylated haemoglobin | -1.3 (1.1) | -1.2 (1.0)

2. Secondary Outcome: Number of Severe and Minor Treatment Emergent Hypoglycaemic Episodes
Description: Confirmed hypoglycaemic episodes consisted of episodes of severe hypoglycaemia as well as minor hypoglycaemic episodes with a confirmed PG value of less than 3.1 mmol/L (56 mg/dL).Minor hypoglycaemic episode is defined as an episode with symptoms consistent with hypoglycaemia with confirmation by full blood glucose < 2.8 mmol/L (50 mg/dL), or PG < 3.1 mmol/L (56 mg/dL) and which is handled by the subject himself/herself or any asymptomatic full blood glucose value < 2.8 mmol/L (50 mg/dL) or PG value < 3.1 mmol/L (56 mg/dL).
Time Frame: On or after the first day of exposure to randomised trial drug (week 0) and no later than 7 days after last exposure to randomised trial drug (week 27)
Population: The Safety analysis set (SAS) included all subjects receiving at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 553 | 278
Episodes/100 years of patient exposure | 85 | 97

3. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose) (Analysed by Central Laboratory)
Description: Change from baseline in FPG after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects. LOCF values are presented for this endpoint. 7 subjects were not included in the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 549 | 277
mmol/L | -3.35 (2.91) | -3.14 (2.71)

4. Secondary Outcome: Within-subject Variability as Measured by Coefficient of Variation (CV%) in Pre-breakfast SMPG (Self-measured Plasma Glucose)
Description: Within subject Coefficient of variation(CV[%]) in pre-breakfast self measured plasma glucose for dose adjustment after 26 treatment weeks are displayed below.
Time Frame: Week 26
Population: The FAS included all randomised subjects. Missing data were imputed using LOCF. For 2 subjects in the IDeg OD arm it was not possible to estimate CV(%) due to missing data.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 553 | 278
percentage | 10.65 (9.15) | 10.01 (7.95)

5. Secondary Outcome: Responder for HbA1c (Below 7.0%) at End of Trial Without Severe and Minor Hypoglycaemic Episodes
Description: A responder for HbA1c without severe or confirmed hypoglycaemia is defined as a subject, who meets the HbA1c target at end of trial without treatment emergent severe or confirmed hypoglycaemia during the last 12 weeks of treatment or within 7 days from last treatment.
Time Frame: Week 26
Population: The FAS included all randomised subjects.
Measure: Number; unit: participants
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 555 | 278
participants | 252 | 114

6. Secondary Outcome: Number of Treatment Emergent AEs (Adverse Events)
Description: Treatment emergent events (after first trial product administration and no later than 7 days after last trial product administration)
Time Frame: On or after the first day of exposure to randomised trial drug (week 0) and no later than seven days after last exposure to randomised trial drug (week 27)
Population: The SAS included all subjects receiving at least one dose of investigational product.
Measure: Number; unit: number of events
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 553 | 278
number of events | 612 | 387

ADVERSE EVENTS:
Time Frame: Treatment emergent events (after first trial product administration and no later than 7 days after last trial product administration)
Description: Safety Analysis Set (SAS) included all subjects receiving at least one dose of investigational product.
Arm/Group | IDeg OD | IGlar OD
Serious Adverse Events (participants affected / at risk) | 16/553 | 10/278
Other Adverse Events (participants affected / at risk) | 100/553 | 58/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=553) | IGlar OD (N=278)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=553) | IGlar OD (N=278)
Nasopharyngitis (Infections and infestations) | 41 (49) | 27 (40)
Upper respiratory tract infection (Infections and infestations) | 60 (77) | 32 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of plans by any investigator to publish and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to Novo Nordisk before submission for comments. Comments will be given within four weeks from receipt of the planned communication.